CLINICAL TRIAL: NCT07345013
Title: A Retrospective Study to Evaluate the Safety and Effectiveness of easyEndoTM Lite Staplers and Loading Units
Brief Title: easyEndoTM Lite Staplers and Loading Units in Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ezisurg Medical Co. Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESM-MDR-VIII 1006A
Record Dates: First submitted 2025-12-17; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Thoracic Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- easyEndoTM Lite linear cutting stapler and loading units (Experimental)
  Interventions: Device: easyEndoTM Lite linear cutting stapler and loading units

INTERVENTIONS:
Device: easyEndoTM Lite linear cutting stapler and loading units — using the easyEndoTM Lite linear cutting stapler and loading units during thoracic surgery

SUMMARY:
A retrospective, single-arm, observation study to Evaluate the clinical safety and performance of Ezisurg stapler in thoracic surgery, 900 patients using the easyEndoTM Lite linear cutting stapler and loading units during thoracic surgery from 2021.03-2022.12 in Fujian Medical University Union Hospital. The surgical decision was made by the surgeons, and no other specification restrictions.

ELIGIBILITY:
The study population were patients using the easyEndoTM Lite linear cutting stapler and loading units during thoracic surgery from 2021.03-2022.12 in Fujian Medical University Union Hospital. The surgical decision was made by the surgeons, and no other specification restrictions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2021-01-03 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
stapling success rate | Perioperative/Periprocedural
  No intrate-operative and post-operative air-leak

SECONDARY OUTCOMES:
Intraoperative blood loss | Perioperative/Periprocedural
Rate of convert to open surgery | Perioperative/Periprocedural
Hospitalization time | Perioperative/Periprocedural
Incidence of postoperative complications | Perioperative/Periprocedural
Readmission rate | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China